CLINICAL TRIAL: NCT07099001
Title: Establishing Clinical Utility Evidence for a Novel Alzheimer's Disease Blood-Based Biomarker Assay: A QURE Virtual Patient Randomized Controlled Trial
Brief Title: Establishing Clinical Utility Evidence for a Novel Alzheimer's Disease Blood-Based Biomarker Assay
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Qure Healthcare, LLC (Industry)
Collaborators: Beckman Coulter, Inc. (Industry)
Responsible Party: Principal Investigator, Trever Burgon, PhD, Principal Investigator, Qure Healthcare, LLC
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: Pro00083791
Record Dates: First submitted 2025-07-16; First posted 2025-08-01 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Alzheimer Disease (AD); Cognitive Decline
Keywords: Patient Simulation
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: The study will enroll neurologists and dementia specialists practicing in the United States. Participants will be randomly assigned to either control or intervention arms upon enrollment. All eligible and consented participants will complete two rounds of three virtual patient simulations.
  The intervention arm participants will receive educational material about the novel Alzheimer's disease assay after round 1 of data collection. After a waiting period, intervention arm participants will receive the results of the AD assay at the appropriate point in the virtual patient simulation. Control arm participants will not receive results of the AD assay, but will have access to standard of care tools during both rounds of case administration.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Control participants will complete two rounds of three virtual patient cases. In both rounds, control participants will have access to standard of care diagnostic tools. They will not receive the AD assay test results.
- Intervention (Experimental): Intervention participants will complete two rounds of three virtual patient cases. In the first round, intervention participants will have access to standard of care diagnostic tools. They will then receive educational material about a novel AD assay. In the second round, they will automatically receive test results for the novel AD assay in addition to standard of care tools.
  Interventions: Other: Educational materials on the Alzheimer's disease assay; Other: Alzheimer's disease assay results

INTERVENTIONS:
Other: Educational materials on the Alzheimer's disease assay — Between Round 1 and Round 2 virtual patient case administration, Intervention participants will receive educational materials describing the clinical validation and use cases of the Alzheimer's disease assay. These materials will approximate the type of information physicians would receive to introduce them to the Alzheimer's disease assay and may be comprised of a slide deck, fact sheet, sample test report, and/or example case scenarios.
  Arms: Intervention
Other: Alzheimer's disease assay results — Within each of their virtual patient cases in Round 2 of case administration, Intervention participants will receive Alzheimer's disease assay results at the clinically appropriate point for each case.
  Arms: Intervention

SUMMARY:
This is a national-level research study of neurologists and dementia specialists. The purpose of this study is to assess the clinical evaluation and management recommendations made by practicing providers for patient simulations with symptoms of cognitive decline.

DETAILED DESCRIPTION:
QURE Healthcare will recruit a nationwide sample of neurologists and dementia specialists to assess the clinical evaluation and management potential of a novel diagnostic tool. The results of this study are expected to contribute to improved quality of care for patients with symptoms of Alzheimer's disease. Findings from this study will be submitted to a national journal for peer-reviewed publication. This study plans to enroll at least 150 healthcare providers.

This study will evaluate the clinical utility of Alzheimer's disease assay by analyzing improvement in the quality of physician decision-making regarding patients with symptoms of Alzheimer's disease, using a validated patient-simulation-based measurement approach, to achieve the following:

1. Measure variation in clinical decisions among practicing neurologists, specifically in how they detect, measure, and manage Alzheimer's disease in patients with symptoms and/or risk factors of cognitive decline.
2. Determine whether education on the Alzheimer's disease assay with accompanying test results leads to changes in clinical decision-making with regard to follow-up testing (e.g., CSF analysis, PET imaging), diagnostic accuracy, and treatment recommendations.
3. Model whether the use of the Alzheimer's disease assay leads to higher-value and/or lower-cost care decisions (including follow-up testing, diagnostics, and treatment) that can lead to more efficient care.
4. Determine whether the Alzheimer's disease assay results differentially impact treatment decisions for different patient types (use cases).

ELIGIBILITY:
Inclusion Criteria:

* Board-certified in neurology for at least two years (and no more than 35 years
* Average at least 20 hours per week of clinical and patient care duties over the past six months
* Routinely evaluate patients at risk for Alzheimer's disease
* Practicing in the United States
* Able to read English
* Access to the internet
* Not participating in a clinical research study of the AD assay
* Informed, signed, and voluntarily consented to participate in this study

Exclusion Criteria:

* Board-certified in neurology for less than two years
* Board certification in neurology over 35 years ago
* Unable to read English
* Unable to access the internet
* Not practicing in the United States
* Not averaging at least 20 hours per week of clinical or patient care duties over the past six months
* Participating in a clinical research study of the AD assay
* Do not voluntarily consent to participate in this study

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-12-31 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
QURE virtual patient clinical score difference | Up to 12 months
  Difference-in-differences regression analysis between the control and the intervention groups' diagnosis and treatment of symptoms of cognitive decline, as measured by the participants' diagnostic and treatment case scores. In each QURE case, every participants' care recommendations are evaluated against evidence-based care scoring criteria, which can range from 0% to 100% (with higher percentages indicating better outcomes).
Change in follow-up decisions (QURE scored-based) after receiving AD assay results | Up to 12 months
  Assessing changes in follow-up decisions (via QURE case domain scores) among intervention providers after they receive the results of the novel AD assay in the second round of case administration. In each QURE case, every participants' care recommendations are evaluated against evidence-based care scoring criteria, which can range from 0% to 100% (with higher percentages indicating better outcomes).

SECONDARY OUTCOMES:
Variation in QURE virtual patient case baseline scores | Up to 12 months
  Participants completing QURE virtual patients receive scores based upon the quality of care they provide. In each QURE case, every participants' care recommendations are evaluated against evidence-based care scoring criteria, which can range from 0% to 100% (with higher percentages indicating better outcomes). This measure will assess the baseline levels of variation in the care of virtual patients with symptoms of cognitive decline among all participants, including by use case types.
Difference in QURE virtual patient case scores by case type | Up to 12 months
  Difference in the overall quality scores between control and intervention participants. The overall score is calculated as the percent of correct (evidence-based) minus incorrect (low-value) decisions divided by the total number of correct decisions in a QURE virtual patient case. Differences in scores between case types across rounds will be assessed to determine which use cases show the most improvement.

CONTACTS AND LOCATIONS:
Overall Officials: Trever Burgon, PhD, Principal Investigator — QURE Healthcare
Locations (1):
- QURE Healthcare, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No